CLINICAL TRIAL: NCT03346603
Title: Prevalence of Extended Spectrum β-lactamase and Carbapenem-Resistant Gram-Negative Bacteria in Patients With Urinary Tract Infection and Urosepsis Admitted Through Emergency Departments in the United States
Brief Title: Prevalence of Antimicrobial-resistant Pathogens in Patients Admitted for UTIs
Status: Completed | Type: Observational
Sponsor: Olive View-UCLA Education & Research Institute (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); IHMA laboratories (Unknown)
Responsible Party: Principal Investigator, David A. Talan, Professor of Medicine in Residence, Olive View-UCLA Education & Research Institute
Other Study IDs: 1057381
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Urinary Tract Infections; Urosepsis
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: urine culture and susceptibility testing — All patients will have a urine culture and susceptibility test ordered per standard care. Results of tests will identify which patients have antimicrobial-resistant organisms.

SUMMARY:
Between 2013-2014, our study network of U.S. emergency departments, EMERGEncy ID NET, found that the rate of fluoroquinolone-resistant E. coli was 11.7% among all patients, 6.3% in uncomplicated and 19.9% in complicated. ESBL-producing Enterobacteriaceae were found in 7.7% of all cases, 2.6% in uncomplicated and 12.2% in complicated. More recently, Enterobactericeae and gram-negative non fermenting bacteria have started to show resistance to carbapenems (CREs and CR-NF). Patients hospitalized with UTI and urosepsis represent a higher risk population for infections due to multi-drug resistant bacteria and experience serious adverse outcomes, including death. EMERGEncy ID NET will conduct a study to determine the prevalence of ESBL-producing, CREs and CR-NFs among this high risk population of patients admitted for UTI from U.S. emergency departments.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years;
2. Admitted to the hospital through the ED;
3. Primary reason for admission is treatment of UTI with or without sepsis (i.e., ED diagnosis of UTI and/or sepsis); and
4. Provide verbal or written consent to participate in the study or if patient is unable to provide consent (e.g., altered mental status), consent obtained from a legal authorized representative.

Exclusion Criteria:

* patients will be later excluded if :

  1. they are unable to provide a urine specimen for culture; or
  2. their urine culture yields no growth or is contaminated (see definition of positive urine culture below). Note: If participant's urine culture is contaminated but their blood culture is positive for a uropathogen, they will not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the 11 U.S. emergency departments involved in the EMERGEncy ID NET study with a urinary tract infection requiring hospital admission.
  The sites are:
  Bellevue Hospital Center, New York; Brigham and Women's Hospital, Boston, MA; Hennepin County Medical Center, Minneapolis; Johns Hopkins Medical Center, Baltimore; Lewis Katz School of Medicine at Temple University, Philadelphia; Maricopa Medical Center, Phoenix; Oregon Health Sciences University, Portland; Olive View-University of California at Los Angeles Medical Center, Los Angeles; University of New Mexico Health Sciences Center, Albuquerque; University of Mississippi Medical Center, Jackson; University of Missouri-Kansas City, Kansas City.
Sampling Method: Non-Probability Sample
Enrollment: 801 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of ESBL-producing Enterobacteriaceae | 2 years
Prevalence of carbapenem-resistant Enterobacteriaceae (CRE) | 2 years
Prevalence of carbapenem-resistant non fermenting gram negative bacteria | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Olive View-UCLA Medical Center, Sylmar, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Final research data will be shared with interested parties affiliated with research organizations, local and U.S. state health departments, and universities, who are interested in using the data for research purposes. Interested parties must submit a short description of how they plan to use the data to the Principal Investigator for approval. A data-sharing agreement will be required containing conditions for data use, including (1): a commitment to using the data only for research purposes; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroy or return the data after analyses are completed. Upon approval, the database will be shared with the requestor. All shared final research databases will not contain direct or indirect personal identifiers, and subjects will only be discernible by unique study identification numbers. A file containing a data dictionary with descriptions of all database fields will be included.
Supporting Information: Study Protocol, ICF
Time Frame: Approximately one year after main manuscript publication. Data will be available for 15 years.
Access Criteria: Data sharing agreement

REFERENCES:
- [Derived] Talan DA, Takhar SS, Krishnadasan A, Mower WR, Pallin DJ, Garg M, Femling J, Rothman RE, Moore JC, Jones AE, Lovecchio F, Jui J, Steele MT, Stubbs AM, Chiang WK, Moran GJ. Emergence of Extended-Spectrum beta-Lactamase Urinary Tract Infections Among Hospitalized Emergency Department Patients in the United States. Ann Emerg Med. 2021 Jan;77(1):32-43. doi: 10.1016/j.annemergmed.2020.08.022. Epub 2020 Oct 31. PMID 33131912